CLINICAL TRIAL: NCT03373812
Title: Comparison Between Different Surgical Approaches for the Treatment of INVOLUTIONAL PTOSIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Arie Nemet, Professor, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMC17230-17CTIL
Record Dates: First submitted 2017-12-04; First posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Involutional Ptosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anterior approach (Active Comparator): patients having involutional ptosis undergoing anterior approach surgical ptosis repair (Levator advancement)
  Interventions: Procedure: Blepharoptosis repair
- posterior approach (Active Comparator): patients having involutional ptosis undergoing posterior approach surgical ptosis repair (mullerectomy)
  Interventions: Procedure: Blepharoptosis repair

INTERVENTIONS:
Procedure: Blepharoptosis repair — levator advancement or mullerectomy

SUMMARY:
Involutional ptosis is a known eyelid pathology in which the eyelid margin obscures part of the visual axis (MRD1).Patients usually complains of visual field disturbance, deterioration in quality of life and a poor cosmetic appearance.

In clinical practice, two main surgical approaches are performed to the repair of involutional ptosis:

1. anterior approach - skin incision and levator muscle insertion advancement.
2. posterior approach - eyelid reversion and tarsectomy Both approaches has its pro's and con's, but to this date, no solid evidence exists to prove which of these techniques is superior in manner of anatomical and functional results.

in this prospective study, patients with involutional ptosis will be randomized to each of surgical approaches groups, parameters concerning surgical and post surgical periods will be evaluated.

DETAILED DESCRIPTION:
Involutional ptosis is a known eyelid pathology in which the eyelid margin obscures part of the visual axis (MRD1).Patients usually complains of visual field disturbance, deterioration in quality of life and a poor cosmetic appearance.

In clinical practice, two main surgical approaches are performed to the repair of involutional ptosis:

1. anterior approach - skin incision and levator muscle insertion advancement.
2. posterior approach - eyelid reversion and tarsectomy Both approaches has its pro's and con's, but to this date, no solid evidence exists to prove which of these techniques is superior in manner of anatomical and functional results.

in this prospective study, patients with involutional ptosis will be randomized to each of surgical approaches groups, parameters concerning surgical and post surgical periods will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Involutional ptosis
* No previous eyelid surgery

Exclusion Criteria:

* Previous eyelid surgery or trauma
* Congenital ptosis
* Previous glaucoma filtrartion surgery
* Unwillingness for six months followup

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
MRD1 | 6 months
  Distance in millimeters between corneal light reflex and upper eyelid margin
surgery duration | 3 hours
  Time from first incision to last suture (in minutes)
Levator function | 6 months
  change (in millimeters) in upper eyelid position from downgaze to maximal upgaze

SECONDARY OUTCOMES:
Need for additional eyelid surgery | 6 months
  Any need for oculoplastic additional surgical interventions (Descriptive)
Eyelid or ocular secondary disease | 6 months
  Descriptive

CONTACTS AND LOCATIONS:
Overall Officials: Arie Nemet, Prof. (MD), Principal Investigator — ophthalmology depertmant, MeirMc, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel RM, Aakalu VK, Setabutr P, Putterman AM. Efficacy of Muller's Muscle and Conjunctiva Resection With or Without Tarsectomy for the Treatment of Severe Involutional Blepharoptosis. Ophthalmic Plast Reconstr Surg. 2017 Jul/Aug;33(4):273-278. doi: 10.1097/IOP.0000000000000748. PMID 27429227
- [Background] Chang S, Lehrman C, Itani K, Rohrich RJ. A systematic review of comparison of upper eyelid involutional ptosis repair techniques: efficacy and complication rates. Plast Reconstr Surg. 2012 Jan;129(1):149-157. doi: 10.1097/PRS.0b013e318230a1c7. PMID 22186506
- [Background] Sohrab MA, Lissner GS. Comparison of Fasanella-Servat and Small-Incision Techniques for Involutional Ptosis Repair. Ophthalmic Plast Reconstr Surg. 2016 Mar-Apr;32(2):98-101. doi: 10.1097/IOP.0000000000000417. PMID 25719375
- [Background] Ben Simon GJ, Joseph J, Lee S, Schwarcz RM, McCann JD, Goldberg RA. External versus endoscopic dacryocystorhinostomy for acquired nasolacrimal duct obstruction in a tertiary referral center. Ophthalmology. 2005 Aug;112(8):1463-8. doi: 10.1016/j.ophtha.2005.03.015. PMID 15953636
- [Background] Liu D. Ptosis repair by single suture aponeurotic tuck. Surgical technique and long-term results. Ophthalmology. 1993 Feb;100(2):251-9. doi: 10.1016/s0161-6420(93)31662-3. PMID 8437835